CLINICAL TRIAL: NCT05739279
Title: Evaluation of Sarcopenia and Associated Factors in Patients with Lipedema
Brief Title: Sarcopenia and Related Factors in Lipedema
Status: Recruiting | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Nihan ERDINC GUNDUZ, Assistant Professor, Dokuz Eylul University
Other Study IDs: 7416-GOA
Record Dates: First submitted 2023-02-12; First posted 2023-02-22 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-08

CONDITIONS: Lipedema; Sarcopenia; Musculoskeletal Diseases
Keywords: Lipedema; Sarcopenia; Musculoskeletal Diseases
MeSH Terms: conditions — Lipedema; Sarcopenia; Musculoskeletal Diseases | interventions — Hand Strength

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Lipedema Group: Patients between the ages of 18-85, diagnosed with lipedema, accepted to participate in the study, and at the appropriate sociocultural level to participate in the study are included in this group.
  Interventions: Diagnostic Test: STAR-Sonographic Thigh Adjustment Ratio; Diagnostic Test: Hand Grip Strength; Diagnostic Test: Chair Stand Test; Diagnostic Test: 6 Meter Gait Speed
- Control Group: Those between the ages of 18-85, in an age group similar to the lipoedema group, who agreed to participate in the study, and who were at the appropriate sociocultural level to participate in the study are included in this group.
  Interventions: Diagnostic Test: STAR-Sonographic Thigh Adjustment Ratio; Diagnostic Test: Hand Grip Strength; Diagnostic Test: Chair Stand Test; Diagnostic Test: 6 Meter Gait Speed

INTERVENTIONS:
Diagnostic Test: STAR-Sonographic Thigh Adjustment Ratio — With ultrasonography, anterior thigh muscle thickness on the dominant extremity side will be measured at a 50% level between the anterior superior iliac spine and the upper pole of the patella in the supine position. The STAR-sonographic thigh adjustment ratio will be calculated by dividing the anterior thigh muscle thickness (mm) by the body mass index.
Diagnostic Test: Hand Grip Strength — Hand grip strength will be measured with a Jamar dynamometer used in the second grip position, in a sitting position with shoulders adducted and neutrally rotated, elbows flexed to 90°, and forearms/wrists in the neutral position. Three repetitive measurements will be made from the dominant side and the maximum value obtained for analysis will be taken.
Diagnostic Test: Chair Stand Test — For the 5-repeat stand-up test, patients will be asked to get up from a chair without an armrest and sit (at the start) five times as fast as possible with their arms crossed over their chest.
Diagnostic Test: 6 Meter Gait Speed — For walking speed measurements, patients will be asked to stand with both feet touching the starting line and walk at their normal speed on a 6-meter track after the command. The time between the start and end will be measured with a stopwatch and converted to meters/second. Three consecutive measurements will be made for both and average values will be taken for the analyses.

SUMMARY:
Lipedema is a common disease of subcutaneous adipose tissue. The most common complaint of patients with swelling in the affected extremity is pain. In addition, patients with lipedema may experience conditions that can greatly affect the health and quality of life of the individual, such as loss of muscle strength and exercise capacity, and deterioration in activity levels of daily living. It is still unknown whether the decrease in muscle strength in patients with lipedema is part of this condition or whether decreased activity levels lead to decreased muscle strength.

Sarcopenia is an important health problem characterized by age-related loss of muscle mass and muscle function. The relationship between muscle weakness and sarcopenia in patients with lipedema has not been investigated before. Early recognition of possible sarcopenia and functional limitations in these patients may be important to increase the ability of patients to participate in physical activity as part of their conservative management.

There is no study in the literature investigating sarcopenia in patients with a diagnosis of lipedema. The aim of this study is to evaluate patients with a diagnosis of lipedema in terms of sarcopenia. In addition, the relationship between sarcopenia and age, body mass index, exercise frequency, lipedema type, and stage will be investigated in patients diagnosed with lipedema.

DETAILED DESCRIPTION:
Lipedema is a chronic progressive condition in women characterized by a disproportionate increase in subcutaneous adipose tissue, accompanied by pain in the legs and sometimes the arms. It was first described in the 1940s and was expressed as fluid accumulation in the wide legs and legs due to subcutaneous fat deposition in the hips and lower extremities. Lipedema is characterized by bilateral enlargement from the hip to the ankle, often sparing the foot, due to abnormal deposition of subcutaneous fat, often with mild edema. The fact that many patients have pain and sensitivity has led to the use of the term painful fat syndrome. The disease usually begins at or just after puberty. Although some lipoedema patients are obese or overweight, the patients often have a normal appearance from the waist up and there is a disproportionate appearance between their trunk and lower extremities. Protection of the hands and feet is typical. This disease, which almost always affects women, has rarely been defined in men due to hormonal disorders or concomitant diseases such as cirrhosis. Although its prevalence is not known exactly, it is thought to be a much more common disease than expected because it is confused with other diseases such as obesity, venous insufficiency, and lymphedema and is a frequently missed diagnosis. Although the results of the studies vary, it has been reported that it is seen at a minimum rate of 1:72.000 or 11% of women affected by this disease.

The pathophysiology of lipoedema is multifactorial, and causes such as increased permeability and capillary fragility due to microangiopathy in adipose tissue, adipocyte necrosis due to hypoxia, and macrophage migration are prioritized. In addition, lymphatic drainage through HIF-1 (hypoxia-inducible factor 1), VEGF (Vascular Endothelial Growth Factor), and FFA (Free Fatty Acid) increases and endothelial barrier function are affected, resulting in impaired vascular circulation due to fluid extravasation and fat accumulation. are held. Estrogen has effects on peripheral and central mechanisms and fat metabolism. The decrease in lipolysis in the femoral region and the increase in lipedema during periods of hormonal changes such as pregnancy, menopause, and oral contraceptive use suggest that hormonal mechanisms are effective on the disease. Preoptic and arcuate nuclei in the hypothalamus; It is involved in lipid mobilization and distribution of white adipose tissue and forms a pathway through ER α (estrogen receptor alpha) and its mediator CART (Cocaine and Amphetamine Regulatory Transcript). Disruption in this regulation pathway also results in regional adipose tissue deposition. There is a family history of 15-64% of the patients, and genetics is thought to be significantly effective. Pedigree studies indicate X-dominant or autosomal-dominant inheritance.

Lipedema usually presents with bilateral extremity swelling that begins in the post-adolescent period, is progressive, does not respond to diet and exercise, does not improve with elevation, and is spontaneous or painful to touch. Patients describe easy bruising with touch or minor trauma. Typically, the hands or feet are not involved, although this may involve the hip and gluteal region. On examination, the skin is often of normal color and texture, and oily hypertrophy may feel soft and pasty. Bruises caused by minor traumas can be observed during the examination. It does not leave pitting after long-term pressure is applied with the finger, and the Stemmer sign, which is observed by compressing the skin on the dorsum of the foot, is negative. Evaluation of these two findings is important in differentiating it from lymphedema. Lipedema consists of 5 major types:

* Type 1 pelvis, gluteal region, and hips,
* Type 2 extending from the gluteal region to the knees and with fat folds in the inner parts of the knees,
* Type 3 extending from the gluteal region to the ankles,
* Type 4 located in arms,
* Type 5 is defined as the presence of isolated swelling in the lower part of the legs.

Types 1-3 are the 3 most common. Lipedema can be seen in 3 stages. In stage 1, the skin surface is normal, the subcutaneous tissue is enlarged, and small nodules are present on palpation. In stage 2, the skin surface is irregular, and large fat nodules are seen. In stage 3, the skin contour is lobulated due to the increase in adipose tissue, and large nodules and deformities are observed. Some sources state the form of lipedema accompanied by lymphedema is stage 4, and this is called lipo lymphedema.

The diagnosis is made clinically, and the history and physical examination can be supported by assistive imaging techniques. The skin and subcutaneous tissue can be examined qualitatively and quantitatively by ultrasonography, computed tomography, or magnetic resonance imaging.

Sarcopenia is an important health problem characterized by age-related loss of muscle mass and muscle function. It is a harbinger of physical fragility and limitation of movement. Muscle wasting is mainly due to the loss of type II muscle fibers, and progressive motor neuron loss is thought to be the primary underlying factor. Anterior thigh muscles atrophy earlier and loss of anterior thigh muscle function may therefore be a precursor finding.

Experts in the sarcopenia special interest group (ISarcoPRM) under the umbrella of the International Society for Physical and Rehabilitation Medicine (ISPRM) have developed a new algorithm based on regional measurements and functional assessments of the anterior thigh muscle, which is initially and most frequently affected in sarcopenia.

The iSarcoPRM has proposed a new measurement that uses anterior thigh muscle measurements for early assessment and rapid diagnosis of low muscle mass and confirmation of sarcopenia. Accordingly, STAR- (sonographic thigh adjustment ratio) sonographic thigh adjustment ratio is found by dividing anterior thigh muscle thickness by body mass index. Using two standard deviation values of healthy young adults, the threshold values for the sonographic thigh fit ratio were found to be 1.4 and 1.0 for male and female subjects, respectively.

As sarcopenia diagnostic criteria;

* STAR- (sonographic thigh adjustment ratio) sonographic thigh adjustment ratio below 1.4 and 1.0 for men and women, respectively
* For muscle strength measurement, hand grip strength is below 32 and 19 kg for men and women, respectively
* It is recommended that the 5-repeat stand-up test (CST (chair stand test)) be longer than 12 seconds.

It has been suggested that walking speed (6 meters) ≤0.8 m/s or inability to get up from a chair without support (limited movement) should be the primary outcome, not part of the diagnostic criteria.

Although pain is the most common complaint of patients with lipoedema along with swelling in the involved extremity, conditions such as loss of muscle strength and exercise capacity, and deterioration in daily life activity levels, can greatly affect the health and quality of life of the individual, can also be seen.

These patients have thickening of the lower extremities beginning in adolescence; limited exercise, dietary changes, or swelling of the affected extremities; they have a medical history that includes limitations in functionality such as fatigue, family history, inability to work, and loss of activity level.

It is still unknown whether the decrease in muscle strength in patients with lipoedema is part of this condition or whether decreased activity levels lead to decreased muscle strength. The relationship between muscle weakness and sarcopenia in these patients has not been investigated before. Early recognition of possible sarcopenia and functional limitations in this patient group may be important to increase the ability of patients to participate in physical activity as a part of conservative management. There is no study in the literature investigating sarcopenia in patients with a diagnosis of lipedema. This study aims to evaluate patients with a diagnosis of lipedema in terms of sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-85
* with a diagnosis of lipoedema
* who agreed to participate in the study
* having a sociocultural level suitable for participation in the study
* healthy volunteers in a similar age group for the control group

Exclusion Criteria:

* with chronic venous insufficiency and/or lymphedema
* with Parkinson's disease, previous stroke, cerebellar diseases, multiple sclerosis, major depression, neuromuscular diseases, history of major orthopedic surgery, severe hip/knee osteoarthritis, rheumatological diseases, malignancies, advanced heart/liver/renal failure, visual impairment, and vestibular diseases, and those who use any assistive device to walk
* who are illiterate and have cognitive impairment that will prevent them from giving written consent will not be included in the study

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Descriptive, cross-sectional, case-control
Sampling Method: Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
STAR-Sonographic Thigh Adjustment Ratio | Day 1
  With ultrasonography, anterior thigh muscle thickness on the dominant extremity side will be measured at a 50% level between the anterior superior iliac spine and the upper pole of the patella in the supine position. The STAR-sonographic thigh adjustment ratio will be calculated by dividing the anterior thigh muscle thickness (mm) by the body mass index.
Hand Grip Strength | Day 1
  Hand grip strength will be measured with a Jamar dynamometer used in the second grip position, in a sitting position with shoulders adducted and neutrally rotated, elbows flexed to 90°, and forearms/wrists in the neutral position. Three repetitive measurements will be made from the dominant side and the maximum value obtained for analysis will be taken.
Chair Stand Test | Day 1
  For the 5-repeat stand-up test, patients will be asked to get up from a chair without an armrest and sit (at the start) five times as fast as possible with their arms crossed over their chest.

SECONDARY OUTCOMES:
6 Meter Gait Speed | Day 1
  For walking speed measurements, patients will be asked to stand with both feet touching the starting line and walk at their normal speed on a 6-meter track after the command. The time between the start and end will be measured with a stopwatch and converted to meters/second. Three consecutive measurements will be made for both and average values will be taken for the analyses

CONTACTS AND LOCATIONS:
Overall Officials: Nihan Erdinc Gunduz, M.D., Study Director — Dokuz Eylul University
Locations (1):
- Department of Physical Medicine and Rehabilitation, Medical Faculty of Dokuz Eylül University, İzmir, Turkey, Izmir, Turkey (Türkiye)